CLINICAL TRIAL: NCT05634759
Title: Enhancing the A in SAFE: Accelerating Trachoma Elimination in the Republic of South Sudan
Brief Title: Enhancing the A in SAFE for Trachoma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Scott Nash, Epidemiologist, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002467
Record Dates: First submitted 2022-11-22; First posted 2022-12-02 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Trachoma
Keywords: Mass drug administration; South Sudan; Trachoma
MeSH Terms: conditions — Trachoma | interventions — Azithromycin

STUDY DESIGN:
Intervention Model Description: Thirty villages will be randomized to one of two intervention arms (15 villages per study arm). To conduct the cost comparison, comparator data for the standard-of-care annual MDA will be obtained from the MDA conducted in 2022 in a random selection of 15 non-study villages.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Routine Community-wide MDA followed by Two Additional Rounds of Treatment for Children (Experimental): The enhanced MDA Strategy 1 consists of a routine community-wide MDA followed by two additional rounds targeted to children age 6 months to 9 years. The additional rounds of treatment will occur 2 weeks apart and will begin 1 week after the community-wide MDA.
  Interventions: Drug: Azithromycin for Routine Community-wide MDA; Drug: Two Additional Rounds of Azithromycin for Children
- Routine Community-wide MDA followed by a Second Community-wide MDA (Experimental): The enhanced MDA Strategy 2 consist of a routine community-wide MDA followed by a second community-wide MDA approximately 6-8 months later. The timing of the second MDA will depend on local conditions and logistical concerns.
  Interventions: Drug: Azithromycin for Routine Community-wide MDA; Drug: Azithromycin for Second Community-wide MDA
- Standard-of-Care Annual MDA (Active Comparator): Programmatic Control Comparator data for the standard-of-care annual MDA will come from the MDA conducted in 2022 in a random selection of 15 non-study villages.
  Interventions: Drug: Azithromycin for Routine Community-wide MDA

INTERVENTIONS:
Drug: Azithromycin for Routine Community-wide MDA — Oral azithromycin, also known as the brand name Zithromax®, is a macrolide antibiotic and is used in the treatment of active trachoma. The recommended dosage for the treatment of trachoma is a single dose of 20mg/kg of body weight and is implemented by a "Age-height" based dosing strategy for the trachoma MDA campaigns. Oral azithromycin can be administrated in either tablet form or powder for oral suspension (POS). Zithromax® is donated by Pfizer Inc through the International Trachoma Initiative (ITI) to the South Sudan Federal Ministry of Health to use in community-wide MDA throughout South Sudan.
  Other Names: Zithromax
Drug: Two Additional Rounds of Azithromycin for Children — An additional round of treatment will be given one week after the routine community-wide MDA, and a second additional round will be given two weeks later (3 weeks after the routine community-wide MDA).
  Other Names: Zithromax
  Arms: Routine Community-wide MDA followed by Two Additional Rounds of Treatment for Children
Drug: Azithromycin for Second Community-wide MDA — A second community-wide MDA will be given 6 to 8 months after the routine community-wide MDA. The timing of the second MDA will depend on local conditions and logistical concerns.
  Other Names: Zithromax
  Arms: Routine Community-wide MDA followed by a Second Community-wide MDA

SUMMARY:
This study will assess the cost and feasibility of two strategies of enhanced Mass Drug Administration (MDA) of Zithromax to treat trachoma in the Republic of South Sudan. The secondary objectives of this study are to measure trachoma infection outcomes during the 12-month follow-up period among children up to 9 years of age.

DETAILED DESCRIPTION:
Trachoma is an ocular disease caused by the bacterium Chlamydia trachomatis. The World Health Organization (WHO) has recently targeted trachoma for global elimination as a public health problem by 2030. Though progress has been made in reducing the burden of trachoma in many endemic countries, those affected by conflict and humanitarian emergencies have been left behind and will likely take decades to reach trachoma elimination targets. To "catch-up", these countries must consider enhancements to the surgery, antibiotic, facial cleanliness, and environmental improvement (SAFE) strategy.

Evidence for the importance of enhanced mass drug administration (MDA) strategies is growing, particularly with the help of modeling studies. Recent work by the neglected tropical disease (NTD) modeling consortium has recently demonstrated that in some hyperendemic districts, annual MDA will not result in a district reaching the elimination as a public health problem threshold within 10 years. Delays in implementation whether due to insecurity or to coronavirus disease 2019 (COVID-19) would likely lead to higher prevalence trachoma prevalence in these districts for years to come. However, when testing alternative MDA strategies, modelers found that the annual trajectory of trachoma prevalence could be changed. One MDA alternative characterized by a community-wide MDA followed by two extra rounds of treatment to children aged 2 to 9 years 1 week and again 3 weeks after the normal community wide MDA, demonstrated a considerable faster time to elimination compared to standard of care. Empirical data from the field under different alternative MDA strategies are needed to verify these modeling results.

The Republic of South Sudan has historically had one of the highest burdens of trachoma in the world. Currently the county has many districts considered highly endemic, and therefore reaching the elimination of trachoma as a public health problem by the year 2030 will likely be a large challenge. Based on 2015 trachoma prevalence data, trachomatous inflammation-follicular among children ages 1 to 9 years ranged from 30% to 48% across three Kapoeta counties in Eastern Equatoria state, Republic of South Sudan and trachomatous trichiasis ranged from 2.6% to 3.7% in those ages 15 years and above, both indicators above WHO elimination thresholds. The Republic of South Sudan Ministry of Health, with support from The Carter Center, has been implementing the SAFE strategy in these three counties (Kapoeta North, Kapoeta South, and Kapoeta East) for over 10 years. Interventions have included the provision of surgery, conducting MDA, and providing health education. All three counties conducted their fifth consecutive annual round of MDA between October 2020 to December 2020 and will therefore be scheduled to conduct an impact survey in 2021.

Thirty villages in the Republic of South Sudan will be randomized to participate in one of two enhanced MDA strategies. Enhanced MDA strategy 1 consists of a routine community-wide MDA followed by two additional rounds targeted to children age 6 months to 9 years. The additional rounds of treatment will occur 2 weeks apart and will begin 1 week after the community-wide MDA. Enhanced MDA Strategy 2 consist of a routine community-wide MDA followed by a second community-wide MDA approximately 6-8 months later. Participants will be followed for 12 months.

ELIGIBILITY:
Inclusion Criteria for Villages:

* The village must be located in a district eligible for annual MDA with azithromycin under WHO treatment guidelines.
* The village representatives' consent to participation in the study. Individual consent will also be obtained for each individual within the study.

Inclusion Criteria for Children in Enhanced MDA Strategy 1:

* Children aged 6 months to 9 years of age
* Consent for child inclusion is obtained by the parent/guardian and adequate provisions are made to solicit assent from the child.

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 34630 (Actual)
Dates: Start 2022-05-04 (Actual); Primary Completion 2023-08-05 (Actual); Study Completion 2023-08-05 (Actual)

PRIMARY OUTCOMES:
Coverage Among Young Children | Up to 12 months
  Feasibility of enhanced antibiotic regimens will be assessed as antibiotic coverage during each of the subsequent treatment rounds, allowing for the calculation of the number of doses each participant received. The definition of coverage for this study is the number of individuals ages 6 months to 9 years who received the drug in study villages in each treatment round divided by number of children ages 6 months to 9 years enumerated in the baseline census. MDA coverage will be further validated through use of the WHO's Supervision Coverage Tool.
Number of Participants Missing Antibiotic Treatment Round | Up to 12 months
  Compliance with the enhanced antibiotic regimens will be assessed as the extent of missed rounds of antibiotic treatment.
Acceptability | Up to 12 months
  The acceptability of enhanced antibiotic regimens will be assessed through focus group discussions which are led by a trained qualitative researcher using a guided discussion tool. Discussion topics include perceptions of trachoma disease and treatment, perception of the MDA campaigns, and community mobilization. This qualitative assessment will not generate a summary score.
Cost | Up to 12 months
  The cost of enhanced antibiotic regimens will be compared to each other and compared to the standard-of-care, annual MDA. The researchers will examine both financial costs (expenditures from the implementation of the intervention), and economic costs (full value of the resources used to implement the intervention). Cost data will be categorized under the following categories: capital costs, medical personnel costs, non-medical personnel costs, commodities, field consumable costs, and lab costs as informed by previous studies.

SECONDARY OUTCOMES:
Prevalence of C. trachomatis Infection | Up to 12 months
  Children age 6 months to 9 years selected for the study will receive ocular swabbing for C. trachomatis infection. The conjunctival epithelial specimen will be used for polymerase chain reaction (PCR) analysis in the lab.
Prevalence of Clinical Trachoma by Field Grader | Up to 12 months
  A field grader will assess both eyes of each child age 6 months to 9 years selected for the study. The grader will note their assessment of trachoma grade prior the ocular swab being obtained.
Prevalence of Clinical Trachoma by Photograph | Up to 12 months
  Tarsal conjunctivae photographs will be taken of both eyes of each child age 6 months to 9 years selected to provide an ocular swab for the study. Images will be sent to a grading center located off-site to be graded by a designated standard grader.
Coverage Among Older Children and Adults | Up to 12 months
  Feasibility of enhanced antibiotic regimens will be assessed as antibiotic coverage during each of the subsequent treatment rounds, allowing for the calculation of the number of doses each participant received. The definition of coverage for this secondary analysis is the number of individuals aged 10 to 15 years, and the number of persons greater than 15 years old who received the drug in study villages in each treatment round divided by number of individuals in each age group enumerated in the baseline census.

OTHER OUTCOMES:
Facial cleanliness | Up to 12 months
  Trained graders will assess facial cleanliness for all children 6 months to 9 years old. The main attributes of facial assessments include presence/lack of ocular and nasal discharge, as well as the time of day of the assessment.
Community awareness of the MDA campaign | Up to 12 months
  A cross-sectional study design will be used to evaluate the impact of the mobilization activities aimed to raise the community's knowledge and awareness of the upcoming MDA campaign.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Nash, PhD, Principal Investigator — The Carter Center
Locations (1):
- Ministry of Health Republic of South Sudan, Juba, South Sudan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sanders AM, Makoy S, Deathe AR, Ohidor S, Jesudason TC, Nute AW, Odongi P, Boniface L, Abuba S, Delahaut AS, Sebit W, Niquette J, Callahan EK, Walker DG, Nash SD. Cost and community acceptability of enhanced antibiotic distribution approaches for trachoma in the Republic of South Sudan: enhancing the A in SAFE (ETAS) study protocol. BMC Ophthalmol. 2023 Feb 6;23(1):51. doi: 10.1186/s12886-023-02783-x. PMID 36747194